CLINICAL TRIAL: NCT02363777
Title: Ultrasound Guided Bilateral Paravertebral Catheters Versus Thoracic Epidural Analgesia for Post- Operative Pain Control in Open Pancreatic Surgery: A Prospective Outcomes Study
Brief Title: Paravertebral Catheters for Pancreatic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1203M11482
Record Dates: First submitted 2015-02-03; First posted 2015-02-16 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Injections, Epidural

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (Active Comparator): Epidural placed for postoperative pain control
  Interventions: Procedure: Epidural
- Experimental Intervention (Experimental): Bilateral paravertebral catheters placed for postoperative pain control
  Interventions: Procedure: Paravertebral catheters

INTERVENTIONS:
Procedure: Epidural — A mid thoracic epidural is placed preoperatively and a local anesthetic and opioid infusion is run postoperatively
  Arms: Standard of Care
Procedure: Paravertebral catheters — Bilateral paravertebral catheters are placed and a local anesthetic infusion via an elastomeric pump is run postoperatively
  Arms: Experimental Intervention

SUMMARY:
Design: Level I randomized prospective outcomes study comparing two groups of patients. One group will receive bupivacaine and dilaudid thoracic epidural analgesia (PCA) post-operatively. The other will receive bilateral ultrasound guided paravertebral blocks with indwelling paravertebral catheters with an infusion of 0.2% ropivicaine post-operatively and a PCA.

Sample Size: 50 patients Study Duration: Approximately 12 months Population:. Patients presenting to the University of Minnesota Medical Center for elective open pancreatic surgery.

Primary Objective: To determine if bilateral paravertebral catheters in patients with open pancreatic procedures result in decreased pain compared to patients treated with thoracic epidural for post-operative pain.

Secondary Objectives:

1. To determine whether the use of bilateral paravertebral catheters impacts the length of ICU and hospital stay for patients, compared to a thoracic epidurals in patients undergoing elective open pancreatic surgery.
2. To determine whether the use of ultrasound guided bilateral paravertebral catheters leads to lower risk of complications, compared to use of a thoracic epidural in patients undergoing open pancreatic surgery.

DETAILED DESCRIPTION:
Design: Level I randomized prospective outcomes study comparing two groups of patients. One group will receive buipvacanine and dilaudid thoracic epidural analgesia (PCA) post-operatively. The other will receive bilateral ultrasound guided paravertebral blocks with indwelling paravertebral catheters with an infusion of 0.2% ropivicaine post-operatively and a PCA.

Sample Size: 50 patients Study Duration: Approximately 12 months Population:. Patients presenting to the University of Minnesota Medical Center for elective open pancreatic surgery.

Primary Objective: To determine if bilateral paravertebral catheters in patients with open pancreatic procedures result in decreased total maximal pain scores compared to patients treated with thoracic epidural for post-operative pain.

Secondary Objectives:

1. To determine whether the use of bilateral paravertebral catheters impacts the length of ICU and hospital stay for patients, compared to a thoracic epidurals in patients undergoing elective open pancreatic surgery.
2. To determine whether the use of ultrasound guided bilateral paravertebral catheters leads to lower risk of complications, compared to use of a thoracic epidural in patients undergoing open pancreatic surgery.

2. Synopsis and Medical Application:

Specific Aims:

Primary Hypothesis: Paravertebral catheters will result in improved pain control relative to thoracic epidural for post-operative pain from open pancreatic surgery.

Secondary Hypothesis: Paravertebral catheters will result in fewer hospital days and improved subjective respiratory function compared to patients in the thoracic epidural group.

ELIGIBILITY:
Inclusion Criteria:

* • All patients undergoing open pancreatic surgery.

Exclusion Criteria:

* • Previous difficult airway or multiple previous intubations

  * History of myasthenic syndrome
  * Systemic infection
  * Pre-existing sensory deficit
  * PT >14 or PTT >40 sec
  * Platelet count less than 50,000
  * Creatinine > 1.5
  * Allergy to local anesthetics
  * Patients who remain intubated for one week after surgery or who are unable to provide information as to their feelings of pain post-operatively for the first week post-operatively
  * Use of a spinal or epidural anesthetic for surgery
  * Daily use of opioid for more than a week or chronic pain syndrome
  * Lack of patient cooperation
  * Contraindication to regional anesthesia

    * Infection at injection site
    * Inability to guarantee sterile equipment or sterile conditions for the block
    * Patient refusal
    * Risk of local anesthetic toxicity
    * Coagulopathy or bleeding disorder
    * Severe respiratory disease (where the patient depends on intercostal muscle function for ventilation);
    * Ipsilateral diaphragmatic paresis;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
total Maximal Pain scored via NRS 0-10 scale | on postoperative day 1 through postoperative day 5
  maximal pain scored via NRS 0-10 scale assessed by independent assessor

SECONDARY OUTCOMES:
Maximal Pain scored via NRS 0-10 scale | on postoperative day 1
  maximal pain scored via NRS 0-10 scale assessed by independent assessor
Maximal Pain scored via NRS 0-10 scale | on postoperative day 2
  maximal pain scored via NRS 0-10 scale assessed by independent assessor
Maximal Pain scored via NRS 0-10 scale | on postoperative day 3
  maximal pain scored via NRS 0-10 scale assessed by independent assessor
Maximal Pain scored via NRS 0-10 scale | on postoperative day 4
  maximal pain scored via NRS 0-10 scale assessed by independent assessor
Maximal Pain scored via NRS 0-10 scale | on postoperative day 5
  maximal pain scored via NRS 0-10 scale assessed by independent assessor
Nausea/vomiting | the first five days postoperatively
  the presence of nausea and or vomiting endorsed by the patient as assessed by an independent assessor
Length of stay | when the patient meets discharge criteria or is discharged home, expected length of stay 10 days
  up through the time the patient is discharged , expected length of stay 10 days.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States